CLINICAL TRIAL: NCT05863845
Title: Efficacy and Safety of Venetoclax Combined With BEAM (Carmustine, Etoposide Cytarabine and Melphalan) Pretreatment in Autologous Stem Cell Transplantation for Diffuse Large B-cell Lymphoma: a Single-center, Randomized Clinical Study
Brief Title: Efficacy and Safety of Venetoclax Combined With BEAM Pretreatment in Autologous Transplantation for DLBCL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Prof., Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V-BEAM
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: LYMPHOMA; DLBCL; ASCT; VENETOCLAX
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — venetoclax; Carmustine; Cytarabine; Etoposide; Melphalan; Stem Cell Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V-BEAM (Experimental): Patients in this arm will receive Venetoclax Combined With BEAM (Carmustine, Etoposide Cytarabine and Melphalan) as Pretreatment Regimen of ASCT.
  Participants receive Venetoclax PO QD on days -10 to -1, Carmustine IV on day -7, Etoposide IV BID on days -6 to -3, Cytarabine IV BID on days -6 to -3, and Melphalan IV on day -2. Participants then undergo hematopoietic cell transplantation on day 0.
  Interventions: Drug: Venetoclax; Drug: Carmustine; Drug: Cytarabine; Drug: Etoposide; Drug: Melphalan; Procedure: Hematopoietic Cell Transplantation
- BEAM (Sham Comparator): Patients in this arm will receive BEAM (Carmustine, Etoposide Cytarabine and Melphalan) as Pretreatment Regimen of ASCT.
  Participants receive Venetoclax PO QD on days -10 to -1, Carmustine IV on day -7, Etoposide IV BID on days -6 to -3, Cytarabine IV BID on days -6 to -3, and Melphalan IV on day -2. Participants then undergo hematopoietic cell transplantation on day 0.
  Interventions: Drug: Carmustine; Drug: Cytarabine; Drug: Etoposide; Drug: Melphalan; Procedure: Hematopoietic Cell Transplantation

INTERVENTIONS:
Drug: Venetoclax — 100mg day -10, 200mg day -9, 400mg day -8, 800mg day -7 to -1, Given PO
  Arms: V-BEAM
Drug: Carmustine — 300mg/m2 day -7, Given IV
Drug: Cytarabine — 100mg/m2/d, day -6 to day -3, Given IV
Drug: Etoposide — 200mg/m2/d, day -6 to day -3, Given IV
Drug: Melphalan — 140mg/m2, day -2, Given IV
Procedure: Hematopoietic Cell Transplantation — Undergo hematopoietic cell transplantation

SUMMARY:
This single-center, randomized clinical study will evaluate the efficacy and safety of Venetoclax combined with BEAM Pretreatment Regimen in ASCT treatment of DLBCL patients.

DETAILED DESCRIPTION:
Diffuse Large B-cell lymphoma (DLBCL) is a group of highly heterogeneous aggressive non-Hodgkin lymphomas with different pathogenesis and clinical prognosis. Despite the survival benefits of Anthracycline-based chemotherapy bridging autologous stem cell transplantation (ASCT), 30%-40% of DLBCL patients fail to respond to treatment and relapse or die within a short period of time. A phase I/II trial of Venetoclax combined with BEAM as a pretreatment regimen for ASCT of high-risk and relapsed/refractory lymphoma was presented at the ASH Meeting 2021 (NCT03583424), and it studies the side effects and best dose of venetoclax when given together with BEAM (carmustine, etoposide, cytarabine, and melphalan) before stem cell transplant in treating participants with relapsed or refractorynon-Hodgkin lymphoma. The results confirmed that Venetoclax has a good prospect in ASCT.

ELIGIBILITY:
Inclusion Criteria:

1. According to world Health Organization (WHO) classification of disease, DLBCL was confirmed by histology, relapsed or refractory after first-line treatment, and CR or PR after upfront treatment;
2. 18≤ age ≤65 years old, male or female;
3. Bcl-2 positive rate >50% according to immunohistochemistry of biopsied tissue;
4. No serious organic lesions in the main organs, meeting the requirements of the following laboratory examination indicators (conducted within 7 days before treatment) :

   * White blood cell count ≥3.0×109/L, absolute neutrophil count ≥1.5×109/L, hemoglobin ≥90g/L, platelet ≥75×109/L;
   * Total bilirubin ≤1.5× upper normal value (ULN);
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5× upper normal value (ULN);
   * Creatinine clearance was 44-133 mmol/L;
5. ECOG score 0-1;
6. The subject or his/her legal representative must provide written informed consent prior to conducting a special study examination or procedure.

Exclusion Criteria:

1. Previously received autologous hematopoietic stem cell transplantation;
2. Suffering from serious complications or severe infection;
3. Previously treated with Venetoclax;
4. Central nervous system lymphoma was excluded; Suffering from serious complications or severe infection;
5. A history of other malignant tumors within 5 years, excluding early tumors treated for curative purposes;
6. Patients with uncontrolled cardiovascular and cerebrovascular diseases, coagulation disorders, connective tissue diseases, serious infectious diseases, etc.;
7. HBsAg, HCV or HIV positive. Positive HBV and HCV serology is allowed, but DNA/RNA testing must be negative;
8. Laboratory test value during screening;

   * Neutrophils <1.5×109/L; Platelet <75×109/L;
   * Bilirubin was 1.5 times higher than the normal upper limit, transaminase was 2.5 times higher than the normal upper limit;
   * The creatinine level is higher than 1.5 times the upper limit of normal value;
9. Left ventricular ejection fraction ≦ 50%;
10. Other concurrent and uncontrolled medical conditions considered by the investigator would affect the patient's participation in the study;
11. Psychiatric patients or other patients known or suspected to be unable to fully comply with the study protocol;
12. Pregnant or lactating women;
13. The researcher judged that the patients were not suitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of ASCT until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from an cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of ASCT to the date of death from any cause.
Complete remission rate | Baseline up to data cut-off (up to approximately 2 years)
  Percentage of participants with complete response was determined on 2014 Lugano criteria.
The time of hematopoietic reconstruction | Baseline up to data cut-off (up to approximately 2 years)
  The first day of neutrophils ≥0.5×109/L for 3 consecutive days was the time of successful implantation of granulocytes. Platelet ≥20.0×109/L for 7 consecutive days and the first day after platelet infusion was considered as the successful time of megakaryocytes implantation.
Transplantation-related adverse reactions | Baseline up to data cut-off (up to approximately 2 years)
  Transplantation-related adverse reactions are any untoward medical occurrence in a participant which is related to ASCT.

IPD SHARING:
Plan to Share IPD: Undecided